CLINICAL TRIAL: NCT06808074
Title: Inhaled Amikacin as a Prophylaxis for Ventilator Associated Pneumonia in Patients With Cirrhosis: A Randomized Placebo Controlled Double Blind Study
Brief Title: A Study to Evaluate Role of Inhaled Amikacin to Prevent Ventilator Associated Pneumonia in Patients With Cirrhosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Anand Kulkarni, Consultant, Department of Hepatology, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AIG/IEC-BH&R 62/09.2024-04
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Encephalopathy; Cirrhosis; Ventilator Associated Pneumonia (VAP)
Keywords: Inhaled amikacin; Prophylaxis; Ventilator associated pneumonia
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaled Amikacin (Experimental)
  Interventions: Drug: Inhaled amikacin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled amikacin — Dosage of amikacin: 20 mg/kg based on ideal body weight, with a maximal dose of 2 g, once daily for 3 consecutive days.
  Arms: Inhaled Amikacin
Drug: Placebo — The equivalent volume of saline solution (0.9% sodium chloride [NaCl]) will be administered once daily for three consecutive days
  Arms: Placebo

SUMMARY:
The recent AMIKINHAL trial found that prophylactic inhaled amikacin was effective in lowering the incidence of ventilator-associated pneumonia in ICU patients. Since aspiration is a common complication of cirrhosis patients with HE (7 out of 10 patients develop some type of HE) who are hospitalized to the liver ICU also have an elevated risk of Ventilator associated pneumonia. Despite supportive care and appropriate antimicrobial therapy pneumonia is linked to greater mortality in cirrhosis. This poses a significant challenge to physicians. Due to the lack of randomized controlled trials (RCTs) on the prophylaxis of VAP in cirrhosis patients with HE, conducting this study is necessary to evaluate the efficacy of inhaled amikacin. The study results may provide evidence -based guidance for therapy in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the liver ICU with hepatic encephalopathy (Grade 2 or higher), requiring intubation for at least 48 hours, without pneumonia.
2. Patient is aged ≥18 years.
3. Written informed consent of the patient or a proxy.

Exclusion Criteria:

1. Suspected or confirmed Pneumonia at the day of inclusion.
2. Patients with Chronic kidney disease on maintenance hemodialysis
3. Stage 2 or 3 Kidney Disease Improving Global Outcome (KDIGO) classification AKI the day of inclusion. Patients undergoing renal replacement therapy or for whom decision has been made to initiate renal replacement therapy can be included whatever the KDIGO stage
4. Pregnancy or breast-feeding.
5. Clinical indication for systemic aminoglycoside therapy the day of inclusion: as deemed necessary by the clinician in charge.
6. Patients known to be allergic to aminoglycosides.
7. Patients who received intravenous Amikacin before 7 days of inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Ventilator associated pneumonia | At day 7 and day 28

SECONDARY OUTCOMES:
All-cause in-hospital mortality | Day 28
Incidence of infections at other sites (Intrabdominal, Blood stream, Urinary tract, Skin and soft tissue) | Day 7, 14, 28
Time to resolution of Hepatic encephalopathy | Day 7, 14, 28
No. of ventilator free ICU days | Day 28
Incidence of Acute kidney injury | Day 7, 14, 28

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - AIG Hospitals, Hyderabad, Telangana
  - Asian Institute of Gastroenterology, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: No